CLINICAL TRIAL: NCT05866796
Title: Validation of Serum GLYcomics to Predict Graft Loss and Mortality After Liver Transplantation
Brief Title: Serum GLYcomics to Predict Graft Loss and Mortality After Liver Transplantation
Acronym: GLYGALT
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: Fund for Scientific Research, Flanders, Belgium (Other); University Hospital, Antwerp (Other); Universitaire Ziekenhuizen KU Leuven (Other); Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2023-0061
Record Dates: First submitted 2023-05-10; First posted 2023-05-19 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Liver Transplant Failure; Prognostic Biomarkers
Keywords: Glycomics; Liver transplantation; Graft survival

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples for glycomics analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No graft loss: Patients receiving liver transplantation that do NOT experience graft loss within 3-months or 12-months after liver transplantation.
  Interventions: Diagnostic Test: GlycoTransplantTest
- Graft loss: Patients receiving liver transplantation that experience graft loss within 3-months or 12-months after liver transplantation.
  Graft loss is defined as either death of the liver transplant recipient (all-cause), or need for retransplantation of the liver.
  Interventions: Diagnostic Test: GlycoTransplantTest

INTERVENTIONS:
Diagnostic Test: GlycoTransplantTest — Determination of serum glycomics in the early posttransplant stage, using an optimal cutoff based on statistic modeling.

SUMMARY:
The first 12 months after liver transplantation (LT) are decisive in posttransplant outcome, as almost half of deaths and two thirds of graft loss requiring retransplant occur in the first year after LT. Since delaying retransplantation in those patients that experience an unfavorable posttransplant course directly impacts their outcome, timely decision making is of paramount importance in these individuals. However, balancing the need and right timing for retransplantation in individual patients with a complicated posttransplant course is currently a difficult challenge that relies on imperfect clinical variables and biomarkers, as well as the experienced judgment of the transplant team.

Building on the findings of a pilot study in liver transplant recipients (n = 131) led by the Ghent University Hospital, we want to validate the prognostic performance of the GlycoTransplantTest on a multicentric scale. In this pilot study, a single glycomic signature at day 7 after LT allowed accurate prediction of graft loss at 3 months after LT. The serum glycome of those patients experiencing graft loss was characterized by increased undergalactosylation and an increased presence of fucosylated and triantennary glycans. After statistical modeling, use of an optimized cutoff based on the relative abundance of 13 serum glycans showed a strong association with graft loss at 3 months (odds ratio 70.211; P<0.001; 95% CI: 10.876-453.23).

Using sequential measurements of serum glycomics in liver transplant recipients, we want to prospectively study and validate the predictive value of the serum glycomic signature for graft survival and overall survival at 3-months (primary end point) and 12-months after liver transplantation (secondary end point).

Determination of the serum glycomic profile is a high-throughput technique that allows to study and quantify the relative abundance of sugar chains (glycans) anchored at specific sites of serum proteins. This technique has shown a very strong prognostic value for graft loss at 3-months after liver transplantation in a pilot study at the Ghent University Hospital.

In this large-scale multicentric prognostic study, we will collect serum samples of liver transplant recipients at fixed time points.

Apart from the serum glycomic profile, we will collect data from the patients electronic record: demographic data (gender, age), data directly relevant to the indication of transplant (eg. imaging for primary liver cancer, lab values for diagnosis of end-stage liver disease), and outcome data (graft survival, overall survival, follow-up time). This list is non-exhaustive.

Using this approach, we will demonstrate the predictive validity of serum glycomics in liver transplant recipients for graft survival and overall survival at 3- and 12-months post-LT. Building on these data, the use of a simple blood test could differentiate patients at risk of graft loss and thus represent a paradigm shift directing these patients to timely treatment adaptations.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated patient informed consent document
* Age ≥ 18 years
* Ability to comply with protocol-specified evaluations and scheduled visits
* Diagnosis of end-stage liver disease, primary hepatic malignancy meeting the Milan criteria for liver transplantation, or acute hepatic failure
* Eligible for liver transplantation and/or active on the waiting list for liver transplantation. Individuals eligible and/or active on the waiting list for multiple organ transplantation including the liver (eg. Combined liver and kidney transplantation, or intestinal transplantation) are also eligible for inclusion.
* Consulted the department of Gastroenterology and Hepatology at Ghent University Hospital

Exclusion Criteria:

- Transplantation of one or more organs not including the liver

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients active on the waiting list or undergoing a liver transplantation. All indications for liver transplantations are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-04-26 (Actual); Primary Completion 2026-04-26 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Graft loss | 3 months after liver transplantation
  Death or need for retransplantation
Mortality | 3 months after liver transplantation
  All-cause mortality

SECONDARY OUTCOMES:
Graft loss | 12 months after liver transplantation
  Death or need for retransplantation
Mortality | 12 months after liver transplantation
  All-cause mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Xavier Verhelst, Ghent, Flanders, Belgium

IPD SHARING:
Plan to Share IPD: Undecided